CLINICAL TRIAL: NCT01676584
Title: A Randomized, Double-blind, Placebo-controlled Single Ascending Dose Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of RO6811135 in Healthy Subjects.
Brief Title: A Study of Single Dose RO6811135 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BP28410
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Healthy Volunteer

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo
- RO6811135 (Experimental)
  Interventions: Drug: RO6811135

INTERVENTIONS:
Drug: RO6811135 — single ascending doses sc
  Arms: RO6811135
Drug: placebo — single doses sc
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled study will evaluate the safety, tolerability, pharmacokinetics and pharmacodynamics of RO6811135 in healthy volunteers. Subjects will be randomized in cohorts to receive either single ascending doses of RO6811135 or placebo subcutaneously.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female volunteers, 18 to 45 years of age inclusive
* Body mass index (BMI) 22-32 kg/m2 inclusive
* Females of child-bearing potential and males with female partners of child-bearing potential must agree to use adequate contraception as defined by protocol

Exclusion Criteria:

* History or presence of any clinically relevant disease or disorder
* History of drug hypersensitivity or food allergies
* Significant infection or known inflammatory process at screening or Day -1
* Any history of alcohol and/or drug of abuse addiction
* Alcohol consumption of more than 14 units (1 unit = 10 mL of pure alcohol) per week
* Smoking more than 5 cigarettes a day or equivalent amount of tobacco
* Positive for hepatitis B, hepatitis C or HIV infection
* Participation in an investigational drug or device study within 3 months prior to screening

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2012-09; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Safety: Incidence of adverse events | approximately 3 months

SECONDARY OUTCOMES:
Pharmacokinetics: Area under the concentration-time curve | Pre-dose and up to 96 hours post-dose
Pharmacodynamics (blood analysis) of RO6811135 | 96 hours

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (1):
- Cincinnati, Ohio, United States